CLINICAL TRIAL: NCT03779776
Title: The Department of Neonatology, Zhengzhou Children's Hospital
Brief Title: The Efficacy and Safety of Early Vitamin AD Supplementation in Very Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou Children's Hospital, China (Other)
Responsible Party: Principal Investigator, Huiqing Sun, Vice Director of Neonatology department, Zhengzhou Children's Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAD-PRETERM
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2020-10

CONDITIONS: Efficacy and Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin AD (Experimental): In Vitamin AD group, the very preterm infants will receive the daily vitamin AD with vitamin A at1500 IU/day and vitamin D at 500 IU/day in drop form added to their enteral feeds when minimal feeding is introduced, and continue to 28 days or discharge. In this group ,the patient also will receive standard intravenous multivitamin preparation (1 ml/kg/d, containing VA 230 IU/kg/d, VD 80 IU/kg/d) within daily on parenteral nutrition until fed 120ml/kg.
  Interventions: Other: Vitamin AD
- Control (Placebo Comparator): In this group ,the patient will only receive standard intravenous multivitamin preparation (1 ml/kg/d,containing VA 230 IU/kg/d,VD 80 IU/kg/d ) within daily on parenteral nutrition until fed 120ml/kg.
  Interventions: Other: Control

INTERVENTIONS:
Other: Vitamin AD — In Vitamin AD group, the very preterm infants will receive the daily vitamin AD with vitamin A at 1500 IU/day and vitamin D at 500 IU/day in drop form added to their enteral feeds when minimal feeding is introduced, and continue to 28 days or discharge. In this group ,the patient also will receive standard intravenous multivitamin preparation (1 ml/kg/d,containing VA 230 IU/kg/d, VD 80 IU/kg/d) within daily on parenteral nutrition until fed 120ml/kg.
  Arms: Vitamin AD
Other: Control — In this group ,the patient will only receive standard intravenous multivitamin preparation (1 ml/kg/d,containing VA 230 IU/kg/d, VD 80 IU/kg/d) within daily on parenteral nutrition until fed 120ml/kg.
  Arms: Control

SUMMARY:
Bronchopulmonary dysplasia (BPD) is the most prevalent longterm morbidity among surviving extremely preterm infants and has a multifactorial etiology. BPD is associated with later risk of reactive airways disease, such as asthma, post neonatal mortality and adverse neurodevelopmental outcomes.Retinopathy of prematurity (ROP) is a common retinal neovascular disorder and a major cause of vision impairment or blindness in preterm infants, even with aggressed current standard care.Accumulating epidemiologic evidence suggests that vitamin D (VD) deficiency or insufficiency is associated with respiratory disease and metabolic bone disease in premature children.Vitamin A (VA) plays an integral part in lung growth and differentiation. VA is an essential micronutrient for normal visual function.

Our prospective double-blinded randomized controlled trial will include infants born at <32 weeks' gestation and admitted to six tertiary NICUs in China. Infants in the intervention (vitamin AD drops) group will receive the daily dose VA at 1500 IU/day with VD 500 IU/day, added to their enteral feeds in drop form as soon as minimal feeding was introduced, and continued to 28 days or discharge. Infants in the control group will receive an equivalent volume of a placebo solution. Following informed consent, enrolled infants will be randomly allocated to the control or VAD group. The primary outcome is bronchopulmonary dysplasia (BPD) , ROP, or metabolic bone disease and the secondary outcomes are mortality; NEC ≥ stage 2; ; late-onset sepsis; weight gain, change in weight, increase in length, increase in head circumference; time to full enteral feeds; and number and type of critical incident reports.

ELIGIBILITY:
Inclusion Criteria:

* gestational age<32 weeks,
* <96 hours of age

Exclusion Criteria:

* genetic metabolic diseases;
* congenital major abnormalities;
* congenital non-bacterial infection with overt signs at birth;
* terminal stage of illness (pH < 7.0 or hypoxia with bradycardia>2 h);
* ≥ grade III intracranial hemorrhage;
* lacking parental consent.

Ages: 1 Hour to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 676 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
rates of bronchopulmonary dysplasia | 1 year
  The rates of bronchopulmonary dysplasia with early vitamin AD supplementation
rates of retinopathy of prematurity | 1 year
  The rates of retinopathy of prematurity with early vitamin AD supplementation
Metaboloc bone disease | 1 year
  The rates of Metaboloc bone disease of prematurity with early vitamin AD supplementation

SECONDARY OUTCOMES:
rates of Necrotizing enterocolitis | 1 year
  The rates of Necrotizing enterocolitis with early vitamin AD supplementation

OTHER OUTCOMES:
rates of late-onset sepsis | 1 year
  The rates of late-onset sepsis with early vitamin AD supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Shuying Luo, MD, Study Director — Zhengzhou Children's Hospital
Locations (1):
- Zhengzhou Children's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No